CLINICAL TRIAL: NCT03985007
Title: Chidamide, Decitabine Combined With Priming IAG Regimen in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: CDIAG Regimen in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, accociate professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZCDIAG
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia, Relapsed, Adult
Keywords: chidamide; decitabine; priming regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CDIAG (Experimental): Relapsed or refractroy acute myeloid leukemia patients reveive chidamide, decitabine combined with priming IAG regimen treatment.
  Interventions: Drug: CDIAG regimen

INTERVENTIONS:
Drug: CDIAG regimen — Chidamide 30mg orally twice every week for 2 weeks on days 1, 4, 8, 11, decitabine 20mg/m2 intravenously daily for 5 days (d1-d5) and IAG regimen (cytarabine, 10 mg/m2 subcutaneously every 12 h on days 4-17; idarubicin, 5mg intravenously every other day on days 4, 6, 8, 10, 12, 14; and concurrent granulocyte colony-stimulating factor, 200mg/m2/day subcutaneously daily on days 3-17.

SUMMARY:
This study is to investigate the therapeutic efficacy and side effect of chidamide, decitabine combined with priming IAG regimen for relapsed or refractroy acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute myeloid leukemia patients without severe complications such as active infections and bleedings; ECOG score less than 3.

Exclusion Criteria:

* Inablity to tolerate inducton chemotherapy; life expectancy less than 1 month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Remission Rate | 1 month
  Remission rate achieved after one-two couses induction therapy by CDIAG regimen
Overall survial | 1 year
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.

SECONDARY OUTCOMES:
Adverse events in hematological system | 1 month
  Record of adverse events in hematological system during and after CDIAG regimen induction
Adverse events in other organs or systems | 1 month
  Record of adverse events in other organs or systmes during and after CDIAG regimen induction

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Yin J, Wan CL, Zhang L, Zhang H, Bai L, Zhou HX, Xu MZ, Chen LY, Qian CS, Qiu HY, Chen SN, Tang XW, Wu DP, Zhang YM, Sun AN, Xue SL. A Phase II Trial of the Double Epigenetic Priming Regimen Including Chidamide and Decitabine for Relapsed/Refractory Acute Myeloid Leukemia. Front Oncol. 2021 Sep 3;11:726926. doi: 10.3389/fonc.2021.726926. eCollection 2021. PMID 34540696